CLINICAL TRIAL: NCT03425708
Title: Study on the Effect of Hyperuricaemia on Chronic Renal Disease and Intervention
Brief Title: Effect of Hyperuricaemia on Chronic Renal Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: The First People's Hospital of Xuzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2017-KL043-01
Record Dates: First submitted 2018-01-13; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Hyperuricemia; Chronic Renal Disease
Keywords: Uric Acid; Febuxostat; Chronic Renal Disease
MeSH Terms: conditions — Hyperuricemia; Renal Insufficiency, Chronic | interventions — Febuxostat; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment group1 (Active Comparator): Febuxostat pill 20mg was used to treat CKD patients with hyperuricaemia.
  Interventions: Drug: 20mg Febuxostat
- Treatment group2 (Active Comparator): Febuxostat pill 40mg was used to treat CKD patients with hyperuricaemia.
  Interventions: Drug: 40mg Febuxostat
- Control group (No Intervention): Treatment of CKD patients with hyperuricaemia with conventional methods.

INTERVENTIONS:
Drug: 20mg Febuxostat — Participants take 20mg febuxostat pill once a day for at least six months.
  Other Names: 20mg Febuxostat pill group
  Arms: Treatment group1
Drug: 40mg Febuxostat — Participants take 40mg febuxostat pill once a day for at least six months.
  Other Names: 40mg Febuxostat pill group
  Arms: Treatment group2

SUMMARY:
To investigate the Effect of Hyperuricaemia on Chronic Renal Disease and Intervention

DETAILED DESCRIPTION:
This study aims to explore the best effective dose and adverse reaction of febuxostat in lowering serum uric acid to low level in patients with Chronic Renal Disease at different stages. To elucidate that low levels of serum uric acid can delay the progression of renal damage. Promote the application of anti uric acid drugs in the treatment of chronic renal failure and delay the progress of CKD in patients

ELIGIBILITY:
Inclusion Criteria:

* Non-dialysis CKD patients with serum uric acid greater than 7mg/dl.
* eGFR≥15ml/min/1.73m².
* Low salt, low protein, low purine diet.

Exclusion Criteria:

* Take drugs that raise blood uric acid at the same time.
* Patients with gout attacks.
* Patients with pregnant, lactating.
* Autosomal dominant polycystic kidney disease.
* Patients with poor general condition and multiple organ failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
serum uric acid | up to 6 months
  intravenous blood sampling

SECONDARY OUTCOMES:
serum creatinine | up to 6 months
  intravenous blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sun, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stack A, Manolis AJ, Ritz E. Detrimental role of hyperuricemia on the cardio-reno-vascular system. Curr Med Res Opin. 2015;31 Suppl 2:21-6. doi: 10.1185/03007995.2015.1087984. PMID 26414733
- [Background] Wang Y, Bao X. Effects of uric acid on endothelial dysfunction in early chronic kidney disease and its mechanisms. Eur J Med Res. 2013 Jul 30;18(1):26. doi: 10.1186/2047-783X-18-26. PMID 23895583 (Retraction: PMID 25890077 Eur J Med Res. 2015;20:44)
- [Background] Tsuruta Y, Kikuchi K, Tsuruta Y, Sasaki Y, Moriyama T, Itabashi M, Takei T, Uchida K, Akiba T, Tsuchiya K, Nitta K. Febuxostat improves endothelial function in hemodialysis patients with hyperuricemia: A randomized controlled study. Hemodial Int. 2015 Oct;19(4):514-20. doi: 10.1111/hdi.12313. Epub 2015 May 21. PMID 25998500
- [Background] Price KL, Sautin YY, Long DA, Zhang L, Miyazaki H, Mu W, Endou H, Johnson RJ. Human vascular smooth muscle cells express a urate transporter. J Am Soc Nephrol. 2006 Jul;17(7):1791-5. doi: 10.1681/ASN.2006030264. Epub 2006 Jun 14. PMID 16775029
- [Background] Khosla UM, Zharikov S, Finch JL, Nakagawa T, Roncal C, Mu W, Krotova K, Block ER, Prabhakar S, Johnson RJ. Hyperuricemia induces endothelial dysfunction. Kidney Int. 2005 May;67(5):1739-42. doi: 10.1111/j.1523-1755.2005.00273.x. PMID 15840020
- [Background] Sellin L, Kielstein JT, de Groot K. [Hyperuricemia - more than gout : Impact on cardiovascular risk and renal insufficiency]. Z Rheumatol. 2015 May;74(4):322-8. doi: 10.1007/s00393-014-1481-1. German. PMID 25962453
- [Background] Mancia G, Grassi G, Borghi C. Hyperuricemia, urate deposition and the association with hypertension. Curr Med Res Opin. 2015;31 Suppl 2:15-9. doi: 10.1185/03007995.2015.1087981. PMID 26414732
- [Background] Miyata H, Takada T, Toyoda Y, Matsuo H, Ichida K, Suzuki H. Identification of Febuxostat as a New Strong ABCG2 Inhibitor: Potential Applications and Risks in Clinical Situations. Front Pharmacol. 2016 Dec 27;7:518. doi: 10.3389/fphar.2016.00518. eCollection 2016. PMID 28082903
- [Background] Perez-Ruiz F, Becker MA. Inflammation: a possible mechanism for a causative role of hyperuricemia/gout in cardiovascular disease. Curr Med Res Opin. 2015;31 Suppl 2:9-14. doi: 10.1185/03007995.2015.1087980. PMID 26414731
- [Background] Tan PK, Ostertag TM, Miner JN. Mechanism of high affinity inhibition of the human urate transporter URAT1. Sci Rep. 2016 Oct 7;6:34995. doi: 10.1038/srep34995. PMID 27713539
- [Background] Sanchez-Lozada LG, Tapia E, Santamaria J, Avila-Casado C, Soto V, Nepomuceno T, Rodriguez-Iturbe B, Johnson RJ, Herrera-Acosta J. Mild hyperuricemia induces vasoconstriction and maintains glomerular hypertension in normal and remnant kidney rats. Kidney Int. 2005 Jan;67(1):237-47. doi: 10.1111/j.1523-1755.2005.00074.x. PMID 15610247
- [Background] Edwards NL. The role of hyperuricemia in vascular disorders. Curr Opin Rheumatol. 2009 Mar;21(2):132-7. doi: 10.1097/BOR.0b013e3283257b96. PMID 19339923
- [Background] Kumagai T, Ota T, Tamura Y, Chang WX, Shibata S, Uchida S. Time to target uric acid to retard CKD progression. Clin Exp Nephrol. 2017 Apr;21(2):182-192. doi: 10.1007/s10157-016-1288-2. Epub 2016 Jun 23. PMID 27339448
- [Background] Srivastava A, Kaze AD, McMullan CJ, Isakova T, Waikar SS. Uric Acid and the Risks of Kidney Failure and Death in Individuals With CKD. Am J Kidney Dis. 2018 Mar;71(3):362-370. doi: 10.1053/j.ajkd.2017.08.017. Epub 2017 Nov 11. PMID 29132945
- [Background] Falvello LR, Fernandez S, Navarro R, Urriolabeitia EP. Reactivity of Pd(0) complexes with the phosphino ylide [Ph2PCH2PPh2=C(H)C(O)Me]. Molecular structure of [Pd(PPh2CHPPh2C(H)C(O)Me)2]. Inorg Chem. 2000 Jun 26;39(13):2957-60. doi: 10.1021/ic990923z. No abstract available. PMID 11232839
- [Background] Kang DH, Ha SK. Uric Acid Puzzle: Dual Role as Anti-oxidantand Pro-oxidant. Electrolyte Blood Press. 2014 Jun;12(1):1-6. doi: 10.5049/EBP.2014.12.1.1. Epub 2014 Jun 30. PMID 25061467
- [Background] Jalal DI, Decker E, Perrenoud L, Nowak KL, Bispham N, Mehta T, Smits G, You Z, Seals D, Chonchol M, Johnson RJ. Vascular Function and Uric Acid-Lowering in Stage 3 CKD. J Am Soc Nephrol. 2017 Mar;28(3):943-952. doi: 10.1681/ASN.2016050521. Epub 2016 Sep 12. PMID 27620990